CLINICAL TRIAL: NCT05643859
Title: Changes in Colonic Microbiome With Fiber Supplementation
Brief Title: Impact of Dietary Fiber Supplementation on Colonic Microbiome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Responsible Party: Principal Investigator, Vassiliki Tsikitis, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00024054; NCI-2022-07495 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00024054 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2022-09-26; First posted 2022-12-09 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Benign Colorectal Neoplasm; Non-Neoplastic Anal Disorder
MeSH Terms: interventions — Dietary Fiber; Proctoscopy; Biopsy; Colonoscopy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive care (oral fiber) (Experimental): Patients receive dietary fiber orally (PO) on study. QD for 28 days. Patients may undergo standard of care proctoscopy or anoscopy with biopsy on study and duringat follow- up or may undergo standard of care colonoscopy on study. All patients also undergo collection of blood samples on study and at follow up.
  Interventions: Dietary Supplement: Dietary Fiber; Procedure: Proctoscopy or anoscopy with Biopsy; Procedure: Colonoscopy; Other: Questionnaire Administration

INTERVENTIONS:
Dietary Supplement: Dietary Fiber — Given PO
  Other Names: Fiber
Procedure: Proctoscopy or anoscopy with Biopsy — Undergo proctoscopy or anoscopy
Procedure: Colonoscopy — Undergo Colonoscopy
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial tests whether daily fiber supplementation will change the mucosal microbiome of the colon. The microbiome are microorganisms that live in the human gut. They serve a vital role in maintaining health. Certain microbial strains are associated with the growth of colon polyps, which eventually could go on to form colon cancer. Giving dietary fiber supplements may help prevent precancerous polyps from ever developing.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To identify how diet, specifically fiber supplementation, alters the microbiome of the colonic mucosa.

OUTLINE:

Patients receive dietary fiber orally (PO) once daily (QD) for 28 days. Patients may undergo standard of care proctoscopy or anoscopy with biopsy on study and at follow up or may undergo standard of care colonoscopy on study. All patients also undergo collection of blood samples on study and at follow up.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Ability to understand and the willingness to sign a written informed consent document
* Patients who present with a chief complaint of a benign anorectal pathology including hemorrhoids, anal fissures, and anal fistulas without underlying conditions such as colorectal cancer or Crohn's disease or are undergoing a standard of care colonoscopy procedure

Exclusion Criteria:

* Patients with an active malignancy, Crohn's disease, ulcerative colitis, and immunosuppressed patients
* Patients with hereditary colon cancer syndrome including Lynch syndrome or Familial Adenomatous Polyposis (FAP)
* Patients with a prior history of total or partial colon resection
* Colorectal pathology, such cancer or proctitis, after initial study scope

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in microbiome colonic mucosa: taxa abundance | Baseline and post-supplementation, up to 40 days
  Will use data visualization techniques to understand the data and determine if microbiome count overall (richness) changes occur in patients who are started on fiber supplementation. In order to visualize overall changes after fiber supplementation, will generate plots showing relative abundance of the detected taxa for each subject at baseline and post-supplementation. For each taxa, will generate box plots to visually compare the median and interquartile range (IQR) of abundance between the two time points. Wilcoxon signed rank tests with an alpha level of 0.05 will determine if there is a difference in microbial derived short chain fatty acids after fiber supplementation in the blood and mucosa. Wilcoxon signed rank tests with an alpha level of 0.05 will determine if there is a difference in microbial derived short chain fatty acids after fiber supplementation in the blood and mucosa.
Change in microbiome colonic mucosa: microbiome diversity | Baseline and post-supplementation, up to 40 days
  Will use data visualization techniques to understand the data and determine if the types of metabolites (microbiome diversity) cases occur in patients who are started on fiber supplementation. In order to visualize overall changes after fiber supplementation. To assess for changes in microbiome diversity, our primary analysis will compare median Shannon diversity index values at baseline and post-supplementation. The Shannon index estimates diversity using richness and abundance. Will calculate Shannon index values for each participant at each time point and use a Wilcoxon signed rank test with an alpha level of 0.05 to determine if there is a difference in microbiome diversity after fiber supplementation.

CONTACTS AND LOCATIONS:
Overall Officials: Vassiliki L Tsikitis, M.D., Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Study team plans to publish the results in the Journal for Microbiome